CLINICAL TRIAL: NCT01298297
Title: Comparison of Sublingual Buprenorphine With Intravenous Morphine Sulfate in Treatment of Acute Pain Due to Long Bone Fracture
Brief Title: Efficacy of Buprenorphine for Treatment of Acute Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUMS-THESIS 88
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Acute Pain
Keywords: Buprenorphine, acute pain, analgesia
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine + Placebo (Active Comparator)
  Interventions: Drug: Buprenorphine
- Morphine + Placebo (Placebo Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Buprenorphine — 0.4 mg, SL (sublingual) Buprenorphine PLUS 5 ml Placebo IV (in the vein)
  Arms: Buprenorphine + Placebo
Drug: Morphine — Placebo SL PLUS 5 ml Morphine sulfate (1mg/ml) IV
  Arms: Morphine + Placebo

SUMMARY:
The purpose of this study is to determine whether sublingual buprenorphine is effective in the treatment of acute pain in adult patients with extremity bone fractures

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of extremity bone fracture Age>16 years Acute pain of score 3 or greater on numerical rating scale

Exclusion Criteria:

Long term use of opium or opioids/dependence Previous administration of analgesic Known sensitivity to opioids Pregnant women History of medical problems (liver, kidney, heart, hematologic)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in pain severity/score | After 60 min

SECONDARY OUTCOMES:
Need for rescue analgesia | After 60 min
Occurrence of adverse events | During 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, Imam Hospital, Tehran, Tehran Province, Iran